CLINICAL TRIAL: NCT03209362
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Repeated Intra-Articular Injection of SI-613 in Patients With Osteoarthritis of the Knee
Brief Title: SI-613 Study for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 613 /1121
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee; Osteoarthritis; Intra-articular injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — diclofenac etalhyaluronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SI-613 (Experimental)
  Interventions: Combination Product: SI-613
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: SI-613 — SI-613 will be repeated intra-articularly administered.
  Arms: SI-613
Combination Product: Placebo — Placebo will be repeated intra-articularly administered.
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of intra-articular injections of SI-613 compared with placebo for knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Provides their written informed consent.
* Has a diagnosis at the time of screening of OA of the knee according to American College of Rheumatology (ACR) criteria
* Is willing to switch to using acetaminophen as a rescue medication

Exclusion Criteria:

* Has a body mass index (BMI) greater than or equal to 40 kg/m2 at screening.
* Secondary OA
* Is a female subject who is pregnant or lactating.
* Is currently hospitalized or has a planned hospitalization during the life of the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - MM Medical Center, Inc., Miami, Florida
  - Quality Research and Medical Center, LLC, Miami, Florida
  - Heartland Research Associates, LLC, Newton, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Rochester Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- SI-613: The participants received repeated intra-articular knee injection of 30 mg SI-613 (1 injection every 4 weeks, total of 3 injections).
- Placebo: The participants received repeated intra-articular knee injection of Placebo (1 injection every 4 weeks, total of 3 injections).
Period: Overall Study
Arm/Group | SI-613 | Placebo
Started | 39 | 41
Completed | 37 | 38
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SI-613 | Placebo | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (7.32) | 59.4 (8.32) | 59.4 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 29
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 34 | 33 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms / meter square] | 30.62 (4.251) | 30.64 (4.669) | 30.63 (4.442)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscore Over 12 Weeks
Description: Observed VAS of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme pain. Change in score from baseline over 12 weeks was analyzed using a repeated measures Analysis of Covariance (ANCOVA) model.
Time Frame: Baseline over 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SI-613 | Placebo
Number analyzed (Participants) | 39 | 41
score on a scale | -29.9 [-36.7 to -23.1] | -27.0 [-33.6 to -20.4]
Statistical Analysis 1: Comparison: SI-613 vs Placebo; Test type: Superiority; p = 0.5453, ANCOVA; Least Squares Mean Difference = -2.9, 95% CI 2-sided [-12.4 to 6.6]

2. Secondary Outcome: Change From Baseline in WOMAC Pain Subscore at Weeks 12 and 26
Description: Observed VAS of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme pain. Changes in score from baseline at Weeks 12 and 26 were analyzed using a longitudinal model.
Time Frame: Baseline, Weeks 12 and 26
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SI-613 | Placebo
Number analyzed (Participants) | 39 | 41
score on a scale
  Change at Week 12 | -40.4 [-48.5 to -32.3] | -36.9 [-44.8 to -28.9]
  Change at Week 26 | -41.7 [-50.2 to -33.1] | -38.4 [-46.7 to -30.1]
Statistical Analysis 1: Comparison: SI-613 vs Placebo; Week 12; Test type: Superiority; p = 0.5386, Longitudinal model; Least Squares Mean Difference = -3.5, 95% CI 2-sided [-14.9 to 7.8]
Statistical Analysis 2: Comparison: SI-613 vs Placebo; Week 26; Test type: Superiority; p = 0.5873, Longitudinal model; Least Squares Mean Difference = -3.3, 95% CI 2-sided [-15.2 to 8.6]

3. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscore at Weeks 12 and 26
Description: Observed VAS of 100 mm; 0 mm meaning no difficulty; 100 mm meaning extreme difficulty. Changes in score from baseline at Weeks 12 and 26 were analyzed using a longitudinal model.
Time Frame: Baseline, Weeks 12 and 26
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SI-613 | Placebo
Number analyzed (Participants) | 39 | 41
score on a scale
  Change at Week 12 | -39.2 [-47.9 to -30.6] | -36.3 [-44.8 to -27.8]
  Change at Week 26 | -38.5 [-47.4 to -29.5] | -36.7 [-45.5 to -28.0]
Statistical Analysis 1: Comparison: SI-613 vs Placebo; Week 12; Test type: Superiority; p = 0.6347, Longitudinal model; Least Squares Mean Difference = -2.9, 95% CI 2-sided [-15.0 to 9.2]
Statistical Analysis 2: Comparison: SI-613 vs Placebo; Week 26; Test type: Superiority; p = 0.7806, Longitudinal model; Least Squares Mean Difference = -1.8, 95% CI 2-sided [-14.3 to 10.8]

4. Secondary Outcome: Change From Baseline in WOMAC Stiffness Subscore at Weeks 12 and 26
Description: Observed VAS of 100 mm; 0 mm meaning no stiffness; 100 mm meaning extreme stiffness. Changes in score from baseline at Weeks 12 and 26 were analyzed using a longitudinal model.
Time Frame: Baseline, Weeks 12 and 26
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SI-613 | Placebo
Number analyzed (Participants) | 39 | 41
score on a scale
  Change at Week 12 | -38.2 [-47.0 to -29.4] | -37.3 [-45.9 to -28.7]
  Change at Week 26 | -41.4 [-50.4 to -32.3] | -35.7 [-44.6 to -26.9]
Statistical Analysis 1: Comparison: SI-613 vs Placebo; Week 12; Test type: Superiority; p = 0.8819, Longitudinal model; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-13.2 to 11.4]
Statistical Analysis 2: Comparison: SI-613 vs Placebo; Week 26; Test type: Superiority; p = 0.3796, Longitudinal model; Least Squares Mean Difference = -5.6, 95% CI 2-sided [-18.3 to 7.1]

5. Secondary Outcome: Change From Baseline in WOMAC Total Score at Weeks 12 and 26
Description: WOMAC total score was the mean of WOMAC pain, physical function and stiffness subscores and ranges from 0 to 100 mm, where higher scores indicated worse response. Changes in WOMAC total score from baseline at Weeks 12 and 26 were analyzed using a longitudinal model.
Time Frame: Baseline, Weeks 12 and 26
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SI-613 | Placebo
Number analyzed (Participants) | 39 | 41
score on a scale
  Change at Week 12 | -39.4 [-47.9 to -30.9] | -36.4 [-44.8 to -28.1]
  Change at Week 26 | -39.4 [-48.2 to -30.6] | -36.9 [-45.5 to -28.3]
Statistical Analysis 1: Comparison: SI-613 vs Placebo; Week 12; Test type: Superiority; p = 0.6217, Longitudinal model; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-14.9 to 9.0]
Statistical Analysis 2: Comparison: SI-613 vs Placebo; Week 26; Test type: Superiority; p = 0.6901, Longitudinal model; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-14.8 to 9.8]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Arm/Group | SI-613 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/41
Other Adverse Events (participants affected / at risk) | 7/39 | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SI-613 (N=39) | Placebo (N=41)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SI-613 (N=39) | Placebo (N=41)
Injection site joint pain (General disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03209362/Prot_SAP_000.pdf